CLINICAL TRIAL: NCT07124689
Title: Relationship Between Central Sensitization Levels and Treatment Outcomes in Patients Diagnosed With Frozen Shoulder and Undergoing Intra-Articular Injection
Brief Title: Relationship Between Central Sensitization Levels and Treatment Outcomes in Frozen Shoulder Treatment
Status: Completed | Type: Observational
Sponsor: Sultan 1. Murat State Hospital (Other Government)
Responsible Party: Principal Investigator, Alper Mengi, Associate Professor, Sultan 1. Murat State Hospital
Other Study IDs: 26/06/2025-Number:37
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Frozen Shoulder; Central Sensitisation; Treatment; Intra-Articular Injection; Shoulder Pain
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Treatment Outcome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with central sensitization: Patients with a score of 40 or higher on theCentral Sensitization Inventory
  Interventions: Other: Treatment outcome
- Patients without central sensitization: Patients with a score below 40 on the Central Sensitization Inventory
  Interventions: Other: Treatment outcome

INTERVENTIONS:
Other: Treatment outcome — Patients will be evaluated for their central sensitization scores before the injection, the pain they experienced during the injection 1 hour after the injection, their daytime and nighttime pain intensity before and 1 month after the injection, their pain thresholds for tactile sensation around the shoulder, and their pain and disability levels.

SUMMARY:
The aim of this study was to evaluate the relationship between treatment outcomes and central sensitization levels in patients who received intra-articular injections for frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 75 years of age
* More than one-third of the active and passive movement of the painful shoulder is limited in two or more planes
* Having pain and limited movement in the shoulder for 3-12 months

Exclusion Criteria:

* Having bilateral shoulder pain
* Patients with incomplete study data
* Having cervical radiculopathy
* Having a predominant central sensitization syndrome (such as fibromyalgia, chronic fatigue syndrome)
* Patients taking antidepressants or anticonvulsants that may affect central sensitization
* Having a history of rheumatological disease
* Having a history of active malignancy
* Patients receiving treatment for active psychiatric disorders
* Having a history of trauma and/or surgery in the same shoulder region
* Patients who received local shoulder injections and/or physical therapy within the last 3 months
* Patients with calcific tendonitis, glenohumeral osteoarthritis, or acromioclavicular joint osteoarthritis on plain radiographs
* Having a full-thickness rotator cuff tear on shoulder ultrasound

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent ultrasound-guided glenohumeral intra-articular injection with a diagnosis of frozen shoulder at Edirne Sultan 1. Murat State Hospital
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2025-08-09 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Presence of Central Sensitization | Baseline
  Patients' levels of central sensitization will be assessed using the Central Sensitization Inventory (CSI). The CSI consists of 25 items, each scored from 0 to 1. A score of 40 or higher indicates the presence of central sensitization.

SECONDARY OUTCOMES:
Post-injection pain severity of patients | Baseline
  Patients will be questioned about their post-injection pain using the Visual Analog Scale (VAS). A 10-cm-long horizontal straight line will be used for VAS assessment. 0 is considered no pain, and 10 is considered the most severe pain.
Patients' daytime pain severity | Baseline
  Patients will be questioned about their daytime pain intensity using the Visual Analog Scale (VAS). A 10-cm-long horizontal straight line will be used for the VAS assessment. 0 is considered no pain, and 10 is considered the most severe pain. Daytime pain intensity will be measured at each assessment as the average pain intensity over the past 48 hours. Daytime pain is measured as the average pain experienced while performing daily routine tasks.
Patients' nighttime pain severity | Baseline
  Patients will be questioned about their nighttime pain intensity using a visual analog scale (VAS). A 10-cm-long horizontal straight line is used for the VAS assessment. 0 is considered no pain, and 10 is considered the most severe pain. Nighttime pain intensity is measured as the average of the pain intensity experienced over the last 48 hours at each assessment. Nighttime pain is questioned as pain upon awakening from sleep or shoulder pain that awakens the patient from sleep.
Pressure pain threshold around the shoulder | Baseline
  Patients' shoulder-area pressure pain thresholds will be assessed using a manual pressure algometer (Baseline Dolorimeter®). Patients' pain perception thresholds will be measured at the midpoint of the bilateral trapezius muscle, the midpoint of the supraspinatus muscle, the midpoint of the deltoid muscle, and the midpoint of the volar aspect of both forearms. During measurement, the 1.52 cm2 flat circular probe of the algometer will be placed on the affected area, and the pressure will be increased at a rate of 1 kg/second. Patients will be asked to report the first time they experience pain. The value for each reference area will be obtained by calculating the arithmetic mean of the paired measurements.
Shoulder-related disability and activities of daily living | Baseline
  Shoulder-related disability and activities of daily living will be assessed using the The Shoulder Pain and Disability Index (SPADI). The SPADI is a 13-item patient completed instrument. Its categories include "pain" (5 items) and "disability" (8 items), with the total score often described as a percentage, resulting from the summation of each component. Overall total scores range from 0 to 130 with a percentage score of 0 indicating less shoulder disability and 100 indicating more shoulder dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan 1. Murat State Hospital, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If requested, the data of the study will be shared by the researchers.